CLINICAL TRIAL: NCT00943813
Title: Assessment of Comskil Training Through Videorecording and Patient Surveys
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-043
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Comskil Training
Keywords: communication; survey; video; 09-043
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients in clinic waiting room: When patients are approached in the clinic, they will be given the permission form and asked to participate in the assessment through allowing video-recording and completing the survey. Procedures will be similar to our current operations, with the RSA starting the video-recording equipment before the fellow enters the room and stopping it when the fellow leaves the room. One additional step will be added: When the RSA goes into the room to turn off and remove the video-recording equipment, she will also give the patient the survey, to complete. We expect this survey to take no longer than 5 minutes. In our experience, it is usually at least 10 minutes from when the fellow leaves the room until the attending comes back into the room. Thus, we believe there will be sufficient time for the patient to complete the survey.
  Interventions: Behavioral: video-recording and completing a survey

INTERVENTIONS:
Behavioral: video-recording and completing a survey — Video record MD consult before MD has completed Comskill training. Post-Video Recording Survey (5 minutes): This is a 22-item self-report scale that measures patient satisfaction and patient reports of communication behavior (Roter et al 1977). Items are rated using a five-point Likert-type scale ranging from 1, "I disagree completely " to 5, "I agree completely ".

SUMMARY:
At Memorial Sloan-Kettering Cancer Center the investigators want to provide the best care to their patients. One way to do this is to evaluate the ways that doctors communicate with patients. To this end, the Department of Psychiatry and Behavioral Sciences runs a Communication Skills Training and Research Laboratory. One goal of this laboratory is to evaluate doctor-patient communication and provide training in how to improve the quality of this communication.

Invitation to participate in this pilot project does not mean that a problem with communication has been identified in your doctor's practice. Rather, it is because your doctor and the fellow working with your doctor have agreed to cooperate with us as the investigators develop strategies to train physicians, nurses and other clinical personnel to communicate with cancer patients in as effective and sensitive a manner as possible.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age;
* Able to understand and provide signature on permission form (Appendix II)
* Able to speak and read English

Exclusion Criteria:

* Evidence of cognitive impairment severe enough to preclude giving permission to the study staff, or completing the survey instrument of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC new visits in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To obtain data from patients about their satisfaction with the fellows' communication and their perception of the fellows' use of communication skills. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bialer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm